CLINICAL TRIAL: NCT02642549
Title: Girls for Health: Empowering Rural Girls' Transition From School to Employment as Health Workers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding
Sponsor: University of California, San Diego (Other)
Collaborators: Center for Girls Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1142975
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Empowerment
MeSH Terms: conditions — Empowerment | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Girls for Health Intervention (G4H) (Experimental): G4H will integrate proven girls' education strategies with innovative vocational interventions to build 1350 girls' career aspirations and academic achievement
  Interventions: Behavioral: Girls for Health
- Control Condition (No Intervention): standard of care to support school attendance among girls (i.e., school tracking of attendance and reaching out to truant girls).

INTERVENTIONS:
Behavioral: Girls for Health — The G4H '1000 Hours' Bridge Program will offer English, science and math training, career workshops, opportunity to 'shadow' a health provider, a mentored safe space club to facilitate economic empowerment, training on gender equity and human rights, and communication/leadership skills. Cash transfers for vacations will be provided to support participation. Girls who receive 5 credits on their SSCE exams and pass the health training institute (HTI) entrance exam are eligible for admission. A Foundational Science Training (FST) program will be provided to the '1000 Hours' participants who gain admission to a HTI to strengthen their ability to the pass the HTI "weeding exams." The FST will focus on English, math and science training, and safe spaces for social support development.
  Other Names: G4H
  Arms: Girls for Health Intervention (G4H)

SUMMARY:
Girls for Health (G4H) will promote the economic empowerment, agency, and voice of rural adolescent girls by supporting their transition from secondary school to tertiary training in midwifery, medicine, nursing and other health careers, and in so doing, will address the acute shortage of female health workers in rural Northern Nigeria. G4H will integrate proven girls' education strategies with innovative vocational interventions to build 1350 girls' career aspirations and academic achievement and will significantly increase the number of rural girls entering health training institutions (HTI) in four northern states. The program will include: 1) a bridge program offering accelerated academic instruction in science, math and English; 2) vocational counseling and practicums at local health facilities; 3) safe spaces to enhance critical life skills; 4) four month science immersion courses for girls accepted for admission to a health training institution; and 5) HTI capacity building to cultivate a rural female-friendly learning environment. G4H will work towards sustainability from the start by using existing secondary school and HTI infrastructure, and feeding into government rural health worker employment schemes.

G4H will be evaluated using a rigorous cluster randomized controlled trial design, randomizing at the school level to assess its impact on key outcomes of interest that include rural girls' secondary school graduation and subsequent HTI enrollment, retention and completion, as well as delayed marriage and improved agency and voice. Process monitoring and costing analysis will be conducted to support quality implementation and dissemination efforts. The design will ensure that high quality evidence is available to guide the field regarding the effectiveness and costing of in-school bridge programming in broadening rural girls' participation in education and career opportunities in the context of low resource settings characterized by low rates of female participation in education and income generation.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in secondary school at selected study schools, in her final two years of secondary school

Exclusion Criteria:

* low attendance (<60%) at participating schools.

Ages: 15 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
completion of secondary school | within 1 year of enrollment
  ascertained via self-report and secondary school records
participation in a HTI (health training institute) or other professional training program | within 1 year of enrollment
  ascertained via self report and vocational school records
graduation from a HTI (health training institute) or other professional training program | within 2 years of enrollment
  ascertained via self-report and vocational school records

SECONDARY OUTCOMES:
delayed marriage | annual follow up over up to 2 years
  ascertained via self report

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Center for Girls Education, Zaria, Kaduna State
  - Federal University Birnin-Kebbi, Kalgo, Kebbi